CLINICAL TRIAL: NCT05531812
Title: Impact of Graduating to Resilience on Child Development in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Doug Parkerson (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); AVSI Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Doug Parkerson, Senior Research Scientist, Director Path-to-Scale Research, Innovations for Poverty Action
Organization: Innovations for Poverty Action (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IPA-2022-UG; 14649-ECD (Other: Innovations for Poverty Action)
Record Dates: First submitted 2022-08-26; First posted 2022-09-08 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Child Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G2R with individual coaching (Experimental)
  Interventions: Other: G2R with individual coaching
- G2R with group coaching (Experimental)
  Interventions: Other: G2R with group coaching
- Control (No Intervention)

INTERVENTIONS:
Other: G2R with individual coaching — 1. Consumption support in the form of a monthly cash transfer for 12 months, totaling US$280-$320;
  2. A one-time "asset" transfer of US$300 delivered ~7 months into the program;
  3. Enrollment, training, and support to participate in a Village Savings and Loans Association (VSLA) or similar group;
  4. Individual coaching at home from a trained coach using a structured curriculum focused on essential topics, including: child nutrition; infant and young child feeding (IYCF) best practices; Water, Sanitation and Hygiene (WASH) practices and practical solutions; preventative health care; positive parenting and life skills; gender; climate risk mitigation strategies; rights, linkages, and access to services.
  Arms: G2R with individual coaching
Other: G2R with group coaching — 1. Consumption support in the form of a monthly cash transfer for 12 months, totaling US$280-$320;
  2. A one-time "asset" transfer of US$300 delivered ~7 months into the program;
  3. Enrollment, training, and support to participate in a Village Savings and Loans Association (VSLA) or similar group;
  4. Group coaching in a community setting from a trained coach using a structured curriculum focused on essential topics, including: child nutrition; infant and young child feeding (IYCF) best practices; WASH practices and practical solutions; preventative health care; positive parenting and life skills; gender; climate risk mitigation strategies; rights, linkages, and access to services.
  Arms: G2R with group coaching

SUMMARY:
This study is an intervention trial that aims to estimate the impact of the Graduating to Resilience (G2R) program on child development in Uganda. In previous trials, the G2R program has generated large, positive impacts on household assets, consumption, income and food security. The investigators will revisit a sample of households enrolled in a G2R trial conducted in Uganda in 2019-2021 (AEARCTR-0004080) and assess children born during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Child born between April 2019 and June 2020
* Household enrolled in G2R intervention trial

Exclusion Criteria:

* None

Ages: 27 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1515 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Bayley Scale of Infant and Toddler Development version III (BSID-III) cognitive z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  Raw item data will be converted to norm-referenced z-scores using the Bayley-III Scoring Assistant software.
BSID-III language z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  Raw item data will be converted to norm-referenced z-scores using the Bayley-III Scoring Assistant software.
BSID-III motor z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  Raw item data will be converted to norm-referenced z-scores using the Bayley-III Scoring Assistant software.
BSID-III social-emotional z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  Raw item data will be converted to norm-referenced z-scores using the Bayley-III Scoring Assistant software.
BSID-III adaptive behavior z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  Raw item data will be converted to norm-referenced z-scores using the Bayley-III Scoring Assistant software.

SECONDARY OUTCOMES:
Caregiver Reported Early Development Instruments (CREDI) cognitive z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  The CREDI long-form will be administered. Raw item data will be converted to norm-referenced z-scores using the CREDI scoring procedure (Waldman et al. 2021).
CREDI language z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  The CREDI long-form will be administered. Raw item data will be converted to norm-referenced z-scores using the CREDI scoring procedure (Waldman et al. 2021).
CREDI motor z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  The CREDI long-form will be administered. Raw item data will be converted to norm-referenced z-scores using the CREDI scoring procedure (Waldman et al. 2021).
CREDI social-emotional z-score | Assessed once approximately 43 months after launch of the intervention in February 2019
  The CREDI long-form will be administered. Raw item data will be converted to norm-referenced z-scores using the CREDI scoring procedure (Waldman et al. 2021).

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Brune, PhD, Principal Investigator — Northwestern University; Nathanael Goldberg, MPA, Principal Investigator — Innovations for Poverty Action; Dean Karlan, PhD, Principal Investigator — Northwestern University; Christopher Udry, PhD, Principal Investigator — Northwestern University; Peter Rockers, ScD, Principal Investigator — Boston University; Doug Parkerson, MA, Principal Investigator — Innovations for Poverty Action
Locations (1):
- Innovations for Poverty Action Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Study data will be published in a public repository
Supporting Information: Study Protocol
Time Frame: Study data will be published concurrent with the publication of the manuscript describing the study results.
Access Criteria: All interested researchers will be able to access and download study data without restrictions.

REFERENCES:
- [Background] Waldman M, McCoy DC, Seiden J, Cuartas J, CREDI Field Team, Fink G. Validation of motor, cognitive, language, and socio-emotional subscales using the caregiver reported early development instruments: an application of multidimensional item factor analysis. International Journal of Behavioral Development 2021;45(4):368-77

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT05531812/SAP_000.pdf